CLINICAL TRIAL: NCT03328728
Title: A Prospective, Multicenter, Randomized,Controlled Study to Compare the Safety and Performance of Cellular Matrix Device (Combination of Autologous Platelet-rich Plasma and Non-crosslinked Hyaluronic Acid) to Those of Synvisc-One (Crosslinked Hyaluronic Acid) for the Treatment of Mild to Moderate Knee Osteoarthritis
Brief Title: Cellular Matrix Device for the Treatment of Mild to Moderate Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-OA-003
Record Dates: First submitted 2017-10-24; First posted 2017-11-01 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cellular Matrix / A-CP HA Kit (Experimental): One intra-articular injection of a combination of PRP and non-crosslinked HA
  Interventions: Device: Cellular Matrix / A-CP HA Kit
- Synvisc-One (Active Comparator): One intra-articular injection of a crosslinked HA
  Interventions: Device: Synvisc-One

INTERVENTIONS:
Device: Cellular Matrix / A-CP HA Kit — Treatment with a single intra-articular injection in the knee of Cellular Matrix / A-CP HA Kit; Cellular Matrix / A-CP HA Kit is designed for the safe, rapid and extemporaneous preparation of a cellular matrix of autologous PRP combined with HA. The Cellular Matrix / A-CP HA Kit is a single-use medical device including hematology tubes (A-CP HA tube), designed for blood collection and PRP/HA preparation after 5 min centrifugation. This tube contains a non-crosslinked hyaluronic acid (MW 1550 kDa) solution, a gel acting as a cell separator, and a sodium citrate acting as an anticoagulant. During centrifugation, the separator gel moves to form a barrier that separates red blood cells from other blood components. The HA, which migrates to the top of the gradient during centrifugation, can be mixed with PRP in order to give rise to a ready-to-use PRP/HA preparation.
  Arms: Cellular Matrix / A-CP HA Kit
Device: Synvisc-One — Treatment with a single intra-articular injection in the knee of Synvisc-One; Synvisc-One (hylan G-F 20) is a sterile, nonpyrogenic, elastoviscous fluid containing hylans. Hylans are derivatives of hyaluronans (sodium salt of hyaluronic acid). Hylan A has an average molecular weight of 6,000,000 daltons and hylan B is a hydrated gel. Hylan G-F 20 contains hylan A and hylan B (8.0 mg per ml) in buffered physiological sodium chloride solution.
  Arms: Synvisc-One

SUMMARY:
This is a non-inferiority study on 190 patients to evaluate whether a treatment based on the combination of autologous platelet-rich plasma and hyaluronic acid obtained with Cellular Matrix represents a therapeutic advantage to relieve symptoms associated with a mild to moderate knee osteoarthritis (particularly pain on walking) compared to hyaluronic acid only (Synvisc®-One).

DETAILED DESCRIPTION:
Platelet-rich plasma (PRP) is an autologous product prepared from the patient's own blood, representing a powerful source of platelet-derived growth factors, particularly useful in the field of regenerative medicine. The active and sequential secretion of these growth factors induces different cell signaling cascades that activate angiogenesis, cell proliferation, cell differentiation, eventually leading to new matrix synthesis and tissue regeneration.

The potential benefits from the use of PRP for the treatment of cartilage defects rely on a number of studies conducted in validated animal models or in vitro, demonstrating the ability of PRP to stimulate collagen production and proteoglycans synthesis, as well as the proliferation and differentiation of mesenchymal stem cells into chondrocytes. Additionally, an increasing number of clinical studies shows an improvement of symptoms, most especially pain, without any occurrence of serious adverse events.

Hyaluronic acid (HA), as one of the major components of the synovial fluid surrounding the cartilage, assumes an important role in the viscoelastic properties of the articular cartilage, conferring its shock absorbing and lubricating functions.

It was demonstrated that rheological properties of synovial fluid decrease with aging and in patients suffering from osteoarthritis. Nowadays, intra-articular injections of hyaluronic acid represent a well recommended therapeutic option to relieve osteoarthritic symptoms, conferring a mechanical action on joints structures, thus leading to reduced pain and improved joint function Based on these data, it seems reasonable to hypothesize that a combination of both PRP and hyaluronic acid could provide greater benefits compared to the administration of each product alone, as their effects on osteoarthritis improvement are based on different mechanisms of action. In fact, on one side PRP promotes cartilage regeneration, while on the other side the HA acts as 3-dimensional support mesh for PRP, providing optimal release of platelets growth factors, strengthening and extending in time the activity of PRP.

Cellular Matrix/A-CP HA Kit is a medical device manufactured by the Swiss company Regen Lab SA. Cellular Matrix/A-CP HA Kit allows to prepare autologous PRP combined with a non-crosslinked hyaluronic acid in a safe, rapid manner and in a single step. The PRP/HA combination is intended to be injected intra-articularly, in order to relieve osteoarthritic symptoms and to improve joint mobility and function. Therefore, the PRP/HA combination might represent a novel therapeutic option for patient suffering from knee osteoarthritis.

This study will evaluate the effects of a single intra-articular injection of a PRP/HA combination prepared with Cellular Matrix/A-CP HA Kit, compared to those of a intra-articular single injection of a well-recognized hyaluronic acid treatment (Synvisc®-One), to relieve symptoms associated with mild to moderate knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* femorotibial knee osteoarthritis defined according to the American College of Rheumatology (ACR) criteria
* Symptomatic knee osteoarthritis of a unilateral knee, characterized by pain at walking (WOMAC A1 score assessed over the previous 24 hours on a 100-mm Visual Analog Scale (VAS): 50 ≤ WOMAC A1 ≤ 90) or reduced joint function (total WOMAC C score assessed or over the previous 24 hours on a 100-mm VAS: 50 ≤ WOMAC A1 ≤ 90)
* Bilateral knee osteoarthritis is allowed, provided the contralateral knee is characterized by a maximum pain of 30 on a 0 to 100 mm scale and doesn't require systemic analgesic treatment, with the exception of paracetamol up to the maximum dose of 4 g per day
* Radiographic femorotibial knee osteoarthritis (radiograph not older than 3 months) Kellgren & Lawrence grades of II-III
* Outpatient capable of walking 50 meters without assistance
* Signature of the informed consent form
* Capable of understanding the study's imperatives, as well as written instructions
* Capable of filling-out evaluation questionnaires

Exclusion Criteria:

* Radiographic femoro-tibial knee osteoarthritis Kellgren & Lawrence grades of I or IV
* Bilateral knee osteoarthritis, characterized by pain greater than 30 of both knees evaluated on a 0 to 100-mm scale and requiring systemic analgesic treatment or paracetamol greater than 4g/ day
* Viscosupplementation in the past 3 months
* Corticosteroid injection in the past 3 months
* PRP or PRP/HA injection in the past 12 months
* Any surgery of the knee planned during the next 6 months
* Systematic use of corticosteroids (except those that are inhaled) or level III analgesics in the past 3 months and NSAID (non-steroidal anti-inflammatory drugs) during the past month
* Treatment with slow-acting anti-rheumatic drugs (diacerhein, soybean or avocado unsaponifiables, chondroitin sulfate, glucosamine) started in the past 6 months
* History of allergy to hyaluronic acid
* Auto-immune disease (rheumatoid arthritis, lupus)
* Surgery of the affected knee in the past 3 months
* Infection of the affected knee in the past 6 months
* Rheumatologic disorder other than arthritis
* Clinical evidence of local inflammation such as redness or heat of the joint
* Hereditary or acquired hematologic or clotting disorders, such as drepanocytosis, platelet dysfunction, thrombocytopenia (<150'000 platelets/mm3), etc.
* Anemia (Hemoglobin < 10g/dl)
* Anticoagulant treatment (patients under antiaggregant treatment can take part to this study as long as their clotting time (CT) is within the reference value)
* Acute infection
* Malignant disease (especially bone and hematological
* serious disorders (cardiovascular pathology, active gastroduodenal ulcer, digestive hemorrhage)
* Patient with renal impairment (creatinine clearance below 45 ml / min)
* Patient with liver failure, pending or who have recently received a liver transplant
* Pregnancy or breastfeeding or planning pregnancy during the course of the study
* Immunosuppression
* Insulin-dependent diabetic patient
* Participation ongoing or in the past 3 months in another clinical study
* Participation to another osteoarthritis clinical study during the past year
* Patient unable to submit to the constraints of the protocol, including patient whose mental condition does not allow him to understand the nature, objectives and possible consequences of the study
* Any other reason which, in the opinion of the investigator, may interfere with the proper conduct of the study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-07-18 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline pain on walking (Western Ontario & McMaster Universities [WOMAC] A1 of the WOMAC questionaire) at 6 months | 6 months
  For each group, pain on walking will be evaluated using a 100-mm Visual Analog Scale (VAS), where 0= no pain and 100 = extreme pain

SECONDARY OUTCOMES:
Change from Baseline pain on walking at 1 and 3 months | 1 and 3 months
  For each group, pain on walking will be evaluated using a 100-mm Visual Analog Scale (VAS), where 0= no pain and 100 = extreme pain
Change from Baseline overall knee osteoarthritis symptoms at 1, 3 and 6 Months | 1, 3 and 6 months
  For each group, overall knee osteoarthritis will be evaluated using the total WOMAC questionnaire; each item of this questionnaire will be scored using a 100-mm VAS at baseline, Month 1, Month 3, and Month 6. The total WOMAC score will be reported as a summed score of all items of the questionnaire, with 0 is the minimum and 2400 is the maximum.
Change from Baseline pain at 1, 3 and 6 Months | 1, 3 and 6 months
  For each group, pain will be evaluated using the WOMAC A subscale; each item of this subscale will be scored using a 100-mm VAS at baseline, Month 1, Month 3, and Month 6. The total WOMAC A score will be reported as a summed score of all items of this subscale, where 0 = is the minimum (no pain) and 500 is the maximum (extreme pain).
Change from Baseline stiffness at 1, 3 and 6 Months | 1, 3 and 6 months
  For each group, stiffness will be evaluated using the WOMAC B subscale; each item of this subscale will be scored using a 100-mm VAS at baseline, Month 1, Month 3, and Month 6. The total WOMAC B score will be reported as a summed score of all items of this subscale, where 0 = is the minimum (no stiffness) and 200 is the maximum (extreme stiffness).
Change from Baseline physical function at 1, 3 and 6 Months | 1, 3 and 6 months
  For each group, physical function will be evaluated using the WOMAC C subscale; each item of this subscale will be scored using a 100-mm VAS at baseline, Month 1, Month 3, and Month 6. The total WOMAC C score will be reported as a summed score of all items of this subscale, where 0 = is the minimum (no difficulty to perform activities) and 1700 is the maximum (extreme difficulty to perform activities).
Change from Baseline quality of life at all time points | 1, 3 and 6 months
  Quality of life will be assessed using the 36-Item Short Form (SF-36) survey that will be given to patients at each visit throughout the study.
Patient Global Assessment of the treatment received | 1, 3 and 6 months
  Patient Global Assessment will be performed using a 5-point numeric scale at 1, 3 and 6 Months, with 1 = completely dissatisfied, 2= dissatisfied, 3 = no change, 4=satisfied , 5= completely satisfied
Clinician Global Assessment of the treatment received | 1, 3 and 6 months
  Patient Global Assessment will be performed using a 5-point numeric scale at 1, 3 and 6 Months, 1 = completely dissatisfied, 2= dissatisfied, 3 = no change, 4=satisfied , 5= completely satisfied
Percentage of OMERACT-OARSI (Outcome Measure in Rheumatology - Osteoarthitis Research Society International) responders at 1, 3 and 6 Months | 1, 3 and 6 months
Percentage of patients requiring an injection of the combination of PRP/HA prepared with Cellular Matrix / A-CP HA at 6 Months | 6 months
Number of local and systemic side effects throughout the study period | 6 months
Cartilage structure | 6 months
  The cartilage structure will be evaluated on the basis of Magnetic Resonance Imaging (MRI) assays at baseline (before receiving the treatment) and 6 months. Differences on the T1 relaxation time parameter will be evaluated at different time points.
Rescue treatment consumption at 1, 3 and 6 Months | 1, 3 and 6 months
  Consumption of authorized medication to relieve pain, according to the patient's diary

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Adam, MD, Principal Investigator — Clinique Médipôle Garonne
Locations (1):
- Clinique Médipôle garonne, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: Undecided